CLINICAL TRIAL: NCT03619642
Title: Reliability, Validity and Clinical Utility of a Robotic Assessment of Finger Proprioception in Neurological Subjects
Brief Title: Reliability, Validity and Clinical Utility of a Robotic Assessment for Proprioception
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hasselt University (Other)
Collaborators: Jessa Hospital (Other); Revalidatie & MS Centrum Overpelt (Other)
Responsible Party: Principal Investigator, Peter Feys, Principal Investigator, Hasselt University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: proprioception01
Record Dates: First submitted 2017-09-14; First posted 2018-08-08 (Actual); Last update posted 2018-09-13 (Actual); Status verified 2018-09

CONDITIONS: Neurological Diseases or Conditions; Sensory Disorders; Multiple Sclerosis; Stroke
MeSH Terms: conditions — Sensation Disorders; Multiple Sclerosis; Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- persons with Multiple Sclerosis (MS) (Other): 25 persons with MS Persons are tested on proprioception of the interphalangeal joints of teh fingers by means of a robotic device.
  Interventions: Other: Robotic assessment of finger proprioception
- stroke patients (Other): 25 stroke patients Persons are tested on proprioception of the interphalangeal joints of teh fingers by means of a robotic device.
  Interventions: Other: Robotic assessment of finger proprioception
- healthy controls (Other): 50 healthy controls Persons are tested on proprioception of the interphalangeal joints of teh fingers by means of a robotic device.
  Interventions: Other: Robotic assessment of finger proprioception

INTERVENTIONS:
Other: Robotic assessment of finger proprioception — The assessment will be performed using a robotic device specifically designed for the assessment of finger proprioception at the metacarpophalangeal (MCP) joint .

SUMMARY:
The aim of this case-controlled observational cross-sectional study is to investigate the test-retest reliability, validity and clinical utility of a rapid robotic assessment of finger proprioception using a passive gauge position matching tasks in MS and stroke subjects.

Session 1 Informed consent Descriptive measures Session 2 Clinical testing Robotic assessment (3x) Session 3 Clinical testing Robotic assessment (3x)

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria MS subjects

* Age > 18 years
* Diagnosis of MS (McDonald criteria)
* No relapse or relapse-related treatment within the last 3 months prior to the study

Inclusion criteria Stroke subjects

* Age > 18 years
* Diagnosis of stroke (ischemic or hemorrhagic),
* Between 2 weeks and 12 months post-stroke

Exclusion Criteria:

* Complete paralysis of both upper limbs
* Unable to detect any passive movement in hand and fingers
* Unable to place the hand in the robotic devices without any discomfort or pain
* Marked or severe intention tremor (Fahn's tremor rating scale on finger-to-nose test > 3)
* Marked or severe spasticity for finger and elbow flexors or shoulder adductors (Modified Asworth scale >3)
* Other medical conditions interfering with the hand function (peripheral nerve lesion, orthopedic or rheumatoid impairment, pain, edema)
* Severe cognitive or visual deficits interfering with testing and training (e.g. Aphasia, neglect, …)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2017-12-15 (Actual); Primary Completion 2018-05-31 (Actual); Study Completion 2018-05-31 (Actual)

PRIMARY OUTCOMES:
Error | day 2
  The extracted parameter is measured by the robotic device. The MCP angular position measured by the robot and the angle reported on the touchscreen by the subject.
Error | day 3
  The extracted parameter is measured by the robotic device. The MCP angular position measured by the robot and the angle reported on the touchscreen by the subject.

SECONDARY OUTCOMES:
sex | day 1
  man/female
Age | day 1
  age
medication use | day 1
  medication use at time of study
the modified Ashworth scale | day 1
  Spasticity of the upper limb will be evaluated with the modified Ashworth scale
Edinburgh Handedness Inventory | day 1
  Hand Dominance evaluated with Edinburgh Handedness Inventory
Nine Hole Peg test | day 1
  manual dexterity test
Box and block test | day 1
  gross and fine upper limb test
Manual Ability Measure-36 (questionnaire) | day 1
  Patient reported measure for upper limb use in daily life activities
Symbol digit modalities test | day 1
  Cognitive function (Symbol digit modalities test)
25 foot walk test | day 1
  Gait velocity test
Semmens-Weinstein monofilaments | day 1
  Tactile sensitivity in the fingers (Semmens-Weinstein monofilaments)
Semmens-Weinstein monofilaments | day 2
  Tactile sensitivity in the fingers (Semmens-Weinstein monofilaments)
Semmens-Weinstein monofilaments | day 3
  Tactile sensitivity in the fingers (Semmens-Weinstein monofilaments)
Rydel Seiffer Tuning fork | day 1
  Vibration in the upper limb (Rydel Seiffer Tuning fork)
Rydel Seiffer Tuning fork | day 2
  Vibration in the upper limb (Rydel Seiffer Tuning fork)
Rydel Seiffer Tuning fork | day 3
  Vibration in the upper limb (Rydel Seiffer Tuning fork)
The Erasmus MC modification of the Nottingham Sensory Assessment (EmNSA) | day 1
  Sensory function test
The Erasmus MC modification of the Nottingham Sensory Assessment (EmNSA) | day 2
  Sensory function test
The Erasmus MC modification of the Nottingham Sensory Assessment (EmNSA) | day 3
  Sensory function test
The System Usability Scale (SUS) | day 2
  Questionnaire
The System Usability Scale (SUS) | day 3
  questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: peter Feys, prof. dr., Principal Investigator — Hasselt University; Joke Raats, Study Chair — Hasselt University; Ilse Jamers, Study Chair — Hasselt University
Locations (2):
- Belgium (2):
  - Jessa Ziekenhuis, Hasselt
  - Revalidatie & MS Centrum Overpelt, Overpelt